CLINICAL TRIAL: NCT00576602
Title: A Randomized, Open Label Study to Evaluate the Effect of Subcutaneous Mircera, Versus no ESA Therapy, on Hemoglobin Levels in Chronic Kidney Disease Patients With Anemia After Kidney Transplant.
Brief Title: A Study of Subcutaneous Mircera, Versus no Erythropoiesis-Stimulating Agent (ESA) Therapy, in the Treatment of Anemia in Patients With Chronic Kidney Disease After Kidney Transplant
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH21299
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator; Palliative Care

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: Supportive treatment

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Recommended starting dose of 0.6 micrograms/kg sc every 2 weeks
  Arms: 1
Drug: Supportive treatment — As prescribed
  Arms: 2

SUMMARY:
This 2 arm study will assess the efficacy, safety and tolerability of subcutaneous Mircera, versus no ESA therapy, in chronic kidney disease patients with anemia after kidney transplant, not currently treated with ESA. Patients will be randomized to receive a)subcutaneous Mircera at a recommended starting dose of 0.6 micrograms/kg every 2 weeks, switching to monthly treatment at week 16 or b)supportive treatment (eg. iron supplementation) for management of low hemoglobin concentrations. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* kidney transplant >=6 months and <5 years prior to randomization;
* anemia;
* no ESA therapy during 3 months prior to randomization.

Exclusion Criteria:

* requirement for hemodialysis or peritoneal dialysis within 3 months prior to randomization;
* change in Hb concentration >=1.5g/dL during screening period;
* transfusion of red blood cells during 3 months prior to randomization;
* poorly controlled hypertension;
* significant acute or chronic bleeding within 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change in Hb concentration between baseline and efficacy evaluation period (EEP). | Weeks 13-16

SECONDARY OUTCOMES:
Change in Hb concentration, percentage of patients maintaining average Hb concentration within target range, percentage of patients requiring dose adjustments, incidence of RBC transfusions. | Throughout study
SF36 | Weeks 16 and 48
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Belgium (3):
  - Edegem
  - Ghent
  - Leuven
- France (7):
  - Amiens
  - Caen
  - Le Kremlin-Bicêtre
  - Nice
  - Paris
  - Toulouse
  - Tours
- Germany (5):
  - Berlin
  - Frankfurt am Main
  - Kaiserslautern
  - Kiel
  - München
- Bari, Italy
- Spain (3):
  - Barcelona
  - Santander
  - Seville
- London, United Kingdom